CLINICAL TRIAL: NCT04931654
Title: A Phase I/IIa Open-label Dose Escalation and Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of AZD7789, an Anti-PD-1 and Anti-TIM-3 Bispecific Antibody, in Participants With Advanced or Metastatic Solid Tumors.
Brief Title: A Study to Assess the Safety and Efficacy of AZD7789 in Participants With Advanced or Metastatic Solid Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9570C00001; 152970 (Registry Identifier: IND); 2022-502774-17 (Registry Identifier: CTIS); 2021-000036-57 (EudraCT Number)
Record Dates: First submitted 2021-05-26; First posted 2021-06-18 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: Solid tumor; Non-small cell lung cancer; NSCLC; Gastric Cancer; Gastroesophageal Junction Cancer; anti-PD-1/PD-L1; anti-TIM-3
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a FTIH, multicenter, open-label, dose-escalation and dose-expansion study. The study includes 2 parts: Part A Dose Escalation and Part B Dose Expansion. Initially, participants with Stage IIIB to IV NSCLC will be enrolled in the study; additional tumor types may be explored and added in a future amendment to the CSP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation Part A: NSCLC Immuno-oncology (IO) acquired or primary resistance (Experimental): AZD7789 monotherapy
  Interventions: Drug: AZD7789
- Dose Expansion Part B1: NSCLC IO acquired resistance - RP2D level 1 (Experimental): AZD7789 Monotherapy
  Interventions: Drug: AZD7789
- Dose Expansion Part B2: NSCLC IO naive, PD-L1 50% or greater - RP2D level 1 (Experimental): AZD7789 Monotherapy
  Interventions: Drug: AZD7789
- Dose Expansion Part B3: NSCLC IO acquired resistance - RP2D level 2 (Experimental): AZD7789 Monotherapy
  Interventions: Drug: AZD7789
- Dose Expansion Part B4: advanced or metastatic gastric and GEJC IO acquired resistance- RP2D level 1 (Experimental): AZD7789 monotherapy
  Interventions: Drug: AZD7789
- Dose Expansion Part B5: NSCLC IO naive, PD-L1 1-49% - RP2D Level 1 (Experimental): AZD7789 monotherapy
  Interventions: Drug: AZD7789

INTERVENTIONS:
Drug: AZD7789 — anti-PD-1 and anti-TIM-3 bispecific antibody

SUMMARY:
This is a Phase I/IIa study designed to evaluate if experimental anti-PD-1 and anti-TIM-3 bispecific antibody, AZD7789 is safe, tolerable and efficacious in participants with advanced solid tumors.

DETAILED DESCRIPTION:
This first time in patients, open-label, multi-centre study will have AZD7789 administered intravenously (IV) to participants with advanced solid tumors. This study will have 2 parts: Part A which will have dose escalation cohorts and Part B which will have the dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years of age
* Part A Dose-escalation cohorts and Part B Dose-expansion cohorts B1, B2, B3 and B5: Histologically or cytologically documented Stage IIIB to IV non-small cell lung carcinoma (NSCLC) not amenable to curative surgery or radiation.
* Part B Dose-expansion cohort B4: Histologically or cytologically documented advanced or metastatic gastric and gastro-esophageal junction adenocarcinoma (GEJC) not amenable to curative surgery or radiation.
* Must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Provision of archival or fresh tumor tissue sample and/or consent to undergo mandatory on-treatment biopsy for participants enrolled in Part A Dose-escalation
* Provision of archival tumor tissue sample or fresh tissue sample for Part B Dose-expansion cohorts B1, B2, B3 and B5. Provision of fresh tumor tissue sample and consent to undergo mandatory on-treatment biopsy for cohort B4.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Non-pregnant women and willingness of female participants to avoid pregnancy or male participants willing to avoid fathering children through highly effective methods of contraception
* Adequate organ and bone marrow function measured within 28 days prior to first dose
* Part A Dose Escalation Additional Inclusion Criteria:

  * May have squamous or non-squamous NSCLC
  * Must have received at least one prior line of systemic therapy, of which at least one prior line of therapy contained approved anti-PD-1/PD-L1
  * Must have had immune-oncology (IO) acquired or primary resistance
  * PD-L1 expression < 1% or ≥ 1% documented
* Part B Dose Expansion Cohort B1 and B3 Additional Inclusion Criteria:

  * May have squamous or non-squamous NSCLC
  * Must have received at least one prior line of systemic therapy, of which only one prior line of therapy contained approved anti-PD-1/PD-L1
  * Must have had IO acquired resistance
  * PD- L1 expression ≥ 1% documented
* Part B Dose Expansion Cohort B2 and B5 Additional Inclusion Criteria:

  * May have squamous or non-squamous NSCLC
  * Must not have received prior IO therapy in the first-line setting, but may have received one prior treatment regime of platinum-based chemotherapy
  * Cohort B2: PD-L1 expression ≥ 50% documented
  * Cohort B5: PD-L1 expression 1-49% documented
* Part B Dose Expansion Cohort B4 Additional Inclusion Criteria:

  * Must have received at least one but no more than two prior lines of systemic therapy, of which only one prior line of therapy contained an approved anti-PD-1/PD-L1
  * Must have had IO acquired resistance
  * There are no PD-L1 status requirements for this cohort

Exclusion Criteria:

* Patients with sensitizing epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) fusions. Documented test result is mandatory for participants with non-squamous NSCLC histology. For participants with squamous NSCLC histology, testing is mandatory only if the participant is a never-smoker or in the presence of a mixed histology.
* Documented test result for any other known genomic alteration for which a targeted first line therapy is approved per local standard of care (SoC)
* Part B Dose-expansion Cohort B4: documented HER2 amplification (unless a SoC including an anti-HER2 therapy has been received); testing is not mandatory if not required per local guidelines.
* Unresolved toxicities of ≥ Grade 2 from prior therapy
* Any prior ≥ Grade 3 immune-mediated adverse event (imAE) while receiving immunotherapy or any unresolved imAE ≥ Grade 2
* Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy
* Symptomatic central nervous system (CNS) metastasis or leptomeningeal disease
* History of symptomatic and objectively confirmed arterial (including myocardial infarction) or venous thromboembolic event within 6 months prior to the first dose of study intervention, unless participant is on treatment with adequate antithrombotic medication and is considered to be stable by the Investigator.
* History of organ transplant or allogenic haematopoietic stem cell transplant
* Infectious disease exclusions: Active infection including TB, HIV, hepatitis A, chronic or active hepatitis B, chronic or active hepatitis C, active COVID-19 infection
* History of clinically significant arrythmia as judged by the Investigator
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiomyopathy of any etiology, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled diabetes mellitus, unstable angina pectoris, history of myocardial infarction within the past 6 months, serious chronic gastrointestinal conditions associated with diarrhea, active non infectious skin disease. Part B Dose-expansion Cohort B4, medication-resistant ascites requiring drainage in the last 28 days prior the start of AZD7789 and/or the occurrence of active gastro-intestinal bleeding, as judged by the Investigator.
* Active or prior documented autoimmune or inflammatory disorders, including inflammatory bowel disease (eg, colitis or Crohn's disease), diverticulitis (with the exception of diverticulosis), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.. Some exceptions have been specified in the protocol
* Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
* Major surgical procedure within 28 days prior to the first dose of study intervention or still recovering from prior surgery
* Other invasive malignancy within 2 years prior to screening
* Congenital long QT syndrome or history of QT prolongation associated with other medications that cannot be changed or discontinued based on a cardiologist assessment
* Any previous treatment with anti-TIM-3 therapy in any setting is not permitted. For Part A, Cohorts B1 and B3:treatment with investigational therapy prior to initiation of study treatment except where the most recent line of therapy was investigational agents added to approved anti-PD-1/PD-L1 as part of standard care. Investigational agents may be given as prior lines of therapy (other than the most recent line) and as monotherapy. Where investigational agents are the most recent line of therapy, they must be given in combination with approved anti-PD-1/PD-L1. For Part B Dose-expansion Cohort B4: investigational agents, other than investigational immune checkpoint inhibitors or other IO agents, may be given as any prior lines of therapy.
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of study intervention
* Any concurrent chemotherapy, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for noncancer-related conditions is acceptable.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention Note: Participants should not receive live vaccine while receiving study intervention and up to 30 days after the last dose of study intervention
* Radiotherapy treatment to the lung within ≤ 4 weeks of the first dose of AZD7789. Palliative bone radiotherapy is allowed if ≥ 2 weeks prior to the first dose of AZD7789.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AE), serious adverse events (SAE) and immune-mediated AEs (imAE) | From time of Informed Consent to 90 days post last dose of study intervention
  Number of participants with AEs, SAEs, imAEs including AEs leading to discontinuation of study intervention and clinically significant alterations in vital signs, laboratory parameters and ECG results
Number of participants with dose-limiting toxicity (DLT), as defined in the protoocol | From the first patient until the end of the dose escalation period; approximately 18 months.
  A DLT is a toxicity defined by the study protocol that occurs from the first dose of study intervention up to the end of the DLT evaluation period that is assessed as clearly unrelated to the primary disease or intercurrent illness.
Preliminary anti-tumour activity of AZD7789 | From first participant until last participant assessment; a duration of approximately 4 years. Disease assessments will be performed until progression or initiation of another anticancer therapy.
  Objective response rate as defined by RECIST v1.1

SECONDARY OUTCOMES:
Objective response rate | From first participant until last participant assessment; a duration of approximately 4 years. Disease assessments will be performed until progression or initiation of another anticancer therapy.
  Objective response rate as defined by RECIST v1.1
Disease control rate | From first documented response to confirmed progressive disease or death; approximate duration of 4 years.
  The percentage of participants according to RECIST v1.1 with a response or stable disease
Duration of response | From first documented response to confirmed progressive disease or death; approximate duration of 4 years.
  The time from first response according to RECIST v1.1 until progression or death
Progression-free survival | From first dose of study intervention to confirmed progressive disease or death; approximate duration of 4 years.
  The time from first dose of study intervention until the date of objective disease progression or death
Overall survival | From first dose of study intervention to death. Overall survival will be monitored for the duration of the study, which will last approximately 4 years.
  The time from first dose of study intervention until death due to any cause
Pharmacokinetics of AZD7789: Maximum plasma concentration of the study drug (Cmax) | From first dose of study intervention, at predefined intervals throughout the administration of study intervention; approximately 4 years.
  Maximum observed plasma concentration of the study drug.
Immunogenicity of AZD7789 | From first dose of study intervention, at predefined intervals throughout the administration of study intervention. A duration of approximately 4 years.
  The number and percentage of participants who develop detectable anti-drug antibodies (ADA).
Pharmacokinetics of AZD7789: Area Under the concentration-time curve (AUC) | From first dose of study intervention, at predefined intervals throughout the administration of study intervention; approximately 4 years.
  Area under the plasma concentration-time curve.
Pharmacokinetics of AZD7789: Clearance | From first dose of study intervention, at predefined intervals throughout the administration of study intervention; approximately 4 years.
  A pharmacokinetic measurement of the volume of plasma from which the study drug is completely removed per unit time.
Pharmacokinetics of AZD7789: Terminal elimination half-life (t 1/2) | From first dose of study intervention, at predefined intervals throughout the administration of study intervention; approximately 4 years.
  Terminal elimination half life.
Preliminary anti-tumour activity of AZD7789: Changes in circulating tumor DNA (ctDNA) | From first dose of study intervention, at predefined intervals throughout the administration of study intervention; approximately 4 years.
  Changes in ctDNA between baseline and on treatment.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (4):
  - Research Site, Atlanta, Georgia
  - Research Site, Fort Wayne, Indiana
  - Research Site, New York, New York
  - Research Site, Nashville, Tennessee
- Research Site, Toronto, Ontario, Canada
- China (2):
  - Research Site, Beijing
  - Research Site, Guangzhou
- France (3):
  - Research Site, Bordeaux
  - Research Site, Rennes
  - Research Site, Villejuif
- Research Site, Tbilisi, Georgia
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kashiwa
- Research Site, Chisinau, Moldova
- Research Site, Amsterdam, Netherlands
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Karşıyaka

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home